CLINICAL TRIAL: NCT06061185
Title: Multimodal Computed Tomography in Patients With Acute Hemorrhagic Stroke (MCTAHS)
Brief Title: Multimodal Computed Tomography in Patients With Acute Hemorrhagic Stroke
Acronym: MCTAHS
Status: Recruiting | Type: Observational
Sponsor: Xiaolin Chen, MD (Other)
Collaborators: Peking University International Hospital (Other); Zhangzhou Municipal Hospital of Fujian Province (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Santai County People's Hospital (Unknown); Jiujiang No.1 People's Hospital (Unknown); Qin Zhou NO.1 People's Hospital (Unknown); Sichuan Academy of Medical Sciences (Other); Linyi People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Xiaolin Chen, MD, Principal Investigator, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Other Study IDs: KY 2024-007-02
Record Dates: First submitted 2023-09-10; First posted 2023-09-29 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Acute Hemorrhagic Stroke
Keywords: Acute Hemorrhagic Stroke; Multimodal CT; Prognosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Testing populations: All patients with the possibility of acute hemorrhagic stroke and suitable for multimodal CT examination
  Interventions: Device: Multimodal CT

INTERVENTIONS:
Device: Multimodal CT — Non-contrast computed tomography, computed tomography angiography and computed tomography perfusion

SUMMARY:
Acute hemorrhagic stroke is a series of neurosurgical diseases characterized by bleeding with high morbidity and mortality. It accounts for about 20% of all strokes worldwide and mainly includes subtypes such as intracerebral hemorrhage (ICH) and subarachnoid hemorrhage (SAH). Multimodal computed tomography including non-contrast computed tomography, computed tomography angiography and computed tomography perfusion, is of great important in understanding pathophysiological changes, evaluating prognosis and guiding interventions in these diseases.

DETAILED DESCRIPTION:
Study overview: The data of the population in the MACTAHS study will be prospectively collected. The CT strategies for acute hemorrhagic stroke are mainly three categories: non-contrast computed tomography, computed tomography angiography and computed tomography perfusion. Each participants will be followed at least until 1 year after discharge. Finally, investigators will clarify the prognostic value of multimodal CT for patients with acute hemorrhagic stroke.

Sample size: About 10000 patients will be enrolled in this study. All the population will be expected to undergo non-contrast computed tomography, computed tomography angiography and computed tomography perfusion.

Study endpoints: Neurological functional outcomes, delayed ischemia and infarction, recurrent bleeding, cognition and emotional dysfunction, systemic in-hospital systemic complications, rehabilitation and recovery status will be evaluated and follow-up would be completed.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18, ≤ 85 years;
2. presence with hemorrhagic stroke

Exclusion Criteria:

1. with a history of previous history of ischemic/hemorrhagic stroke;
2. admission to the emergency department more than a week after symptom onset;
3. serious medical history or existing comorbidities;
4. physical disability due to previous diseases;
5. prior treatment such as external ventricular drainage, digital subtraction angiography and lumbar puncture in other institution;
6. poor original image quality;
7. incomplete follow-up.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presented to the emergency department with hemorrhagic stroke.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2032-03-01 (Estimated); Study Completion 2032-04-01 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) | At 3/6/12 months after onset
  The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms.
  No significant disability. Able to carry out all usual activities, despite some symptoms.
  Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  Moderate disability. Requires some help, but able to walk unassisted. Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  Dead

SECONDARY OUTCOMES:
Mortality rate | At 12 months after onset
  Mortality rate as measured by death of a participant (binary outcome (yes/no)
Total time spent on the intensive care unit (ICU)/stroke unit | After treatment (max 60 days)
  The total time spent on the intensive care unit (ICU)/stroke unit as a continuous variable from the first admission to the ICU/stroke unit to discharge from ICU/stroke unit
Non-neurological systemic complications | After onset (max 60 days)
  This category of diseases mainly refers to a series of non-neurological systemic complication such as electrolyte alterations, cardiovascular complications, pneumonia, gastrointestinal alterations, coagulation disorders and so on
Delayed infarction | After onset (max 30 days)
  Delayed onset of any type of infarction detected by NCCT/MRI/CTP after surgical treatment or during conservative treatment
Delayed ischemia | After onset (max 30 days)
  Delayed onset of various types of ischemia detected by PWI/CTP after surgical treatment or during conservative treatment, as well as a short period decline of cognitive and neurological status
Hematoma expansion in intracerebral hemorrhage | 24-48 hours from symptom onset
  non-contrast CT scan: the enlargement of hematoma ≥ 6ml
Recurrence of intracerebral hemorrhage | 90 days from symptom onset
  non-contrast CT scan: non-traumatic intracerebral hemorrhage other than the primary bleeding
Rebleeding of subarachnoid hemorrhage | After onset (max 7 days)
  Rebleeding Hemorrhage in subarachnoid space proven on CT/MR scan
Montreal Cognitive Assessment Scale (MoCA) | At 3/6/12 months after onset
  It included 11 tests in eight cognitive areas: attention and concentration, executive function, memory, language, visual structure skills, abstract thinking, computation, and orientation. Total score 30, ≥26 normal
Mini-mental State Examination (MMSE) | At 3/6/12 months after onset
  The scale includes the following seven aspects: time orientation, place orientation, immediate memory, attention and computation, delayed memory, language, visual space. A total of 30 questions, each correct answer is 1 point, the answer is wrong or do not know 0 points, the scale total range of 0-30 points. Test scores are closely related to literacy level, and the normal cut-off values are: illiterate >17 points, primary >20 points, junior high school and above >24 points.
Self-Rating Anxiety Scale (SAS) | At 3/6/12 months after onset
  The scale consists of 20 items with 4 marks for each item. The scores of each of the 20 items are added together, and then multiplied by 1.25 to get the integer part. The total score of anxiety less than 50 points is normal; 50-60 is mild, 61-70 is moderate, and over 70 is severe anxiety.
Self-Rating Depression Scale (SDS) | At 3/6/12 months after onset
  The scale consists of 20 items with 4 marks for each item. The scores of each of the 20 items are added together, and then multiplied by 1.25 to get the integer part. The cut-off value of the SDS standard score is 53 points, of which 53-62 is classified as mild depression, 63-72 is classified as moderate depression, and 73 or more is severe depression.
Hamilton Rating Scale for Anxiety | At 3/6/12 months after onset
  Anxiety will be assessed using the Hamilton Rating Scale for Anxiety. The Hamilton Anxiety Rating Scale measures the severity of anxiety through looking at both psychic and somatic anxiety. Each item is scored on a scale of 0 to 4, with a total range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Hamilton Rating Scale for Depression | At 3/6/12 months after onset
  Depression will be assessed using the Hamilton Rating Scale for Depression (HAM-D). The HAM-D is a 21 item questionnaire to treat and diagnosis severe depression. Examining a different symptom or aspect of depression such as mood, guilty feelings, suicidal ideation, etc.. The first 17 questions are used for scoring. A total score is tallied from 1-17 and if the score totals: 0-7 normal, 8-13 mild depression, 14-18 moderate depression, 19-22 severe depression, >23 very severe depression.
Fatigue | At 12 months after onset
  Fatigue will be assessed using the Fatigue Severity Scale. The Fatigue Severity Scale measures the severity of fatigue and its effect on a person's activities and lifestyle in patients exhibiting depression. The scale is designed to differentiate fatigue from clinical depression since they share similar symptoms. Scoring is done by calculating the average response to the question and people with depression typically score about 4.5 whereas those with fatigue average about 6.5.

CONTACTS AND LOCATIONS:
Overall Officials: Tu Li, M.D., Study Chair — Beijing Tiantan Hospital; Zhenshan Song, M.D., Study Chair — Beijing Tiantan Hospital; Runting Li, M.D., Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided